CLINICAL TRIAL: NCT02719639
Title: Assessment of Physical Functioning and Handling of Spiolto Respimat in Patients With Chronic Obstructive Pulmonary Disease (COPD) Requiring Long-acting Dual Bronchodilation in Routine Clinical Practice.
Brief Title: OTIVACTO Regional Center Vienna (RCV) Non-Interventional Study (NIS)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.44
Record Dates: First submitted 2016-03-01; First posted 2016-03-25 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Real-world data on the effects of a fixed-dose combination Long-acting beta agonists + long-acting antimuscarinic agent (LABA+LAMA) therapy with tiotropium and olodaterol administered in a single device, in COPD patients who need treatment with two long-acting bronchodilators, is not available. This is a self-controlled study design enrolling consented COPD patients who will be treated with Spiolto Respimat according to the approved Summary of Product Characteristics (SmPC).

DETAILED DESCRIPTION:
Purpose:

Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to participation
2. Female and male patients with more or equal to 40 years of age
3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto Respimat Summary of Product Characteristics (SmPC) and chronic obstructive pulmonary disease (COPD) Global Initiative for Chronic Obstructive Lung Disease (GOLD) guideline recommendation

Exclusion criteria:

1. Patients with contraindications according to Spiolto Respimat SmPC
2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months
3. Patients continuing LABA- Inhalative Corticosteroids (ICS) treatment should not be additionally treated with Spiolto Respimat in order to avoid a double dosing of long-acting beta-agonists
4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
5. Pregnancy and lactation
6. Patients currently listed for lung transplantation
7. Current participation in any clinical trial or any other non-interventional study of a drug or device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPDS patients
Sampling Method: Probability Sample
Enrollment: 7443 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- Multiple Locations, Austria
- Multiple Locations, Czechia
- Multiple Locations, Hungary
- Multiple Locations, Israel
- Multiple Locations, Romania
- Multiple Locations, Russia
- Multiple Locations, Slovakia
- Multiple Locations, Slovenia
- Multiple Locations, Switzerland

REFERENCES:
- [Derived] Taube C, Bayer V, Zehendner CM, Valipour A. Assessment of Patient Experiences with Respimat(R) in Everyday Clinical Practice. Pulm Ther. 2020 Dec;6(2):371-380. doi: 10.1007/s41030-020-00127-4. Epub 2020 Aug 28. PMID 32857327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open label observational study in Chronic Obstructive Pulmonary Disease (COPD) patients from 534 investigational sites in 9 countries.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be entered to trial if any one of the specific entry criteria were not met.
Groups:
- Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram: Patients with Chronic Obstructive Pulmonary Disease (COPD) included in this group were treated with Spiolto® Respimat®, Tiotropium/ Olodaterol 2.5 microgram/ 2.5 microgram, inhalation solution for 6 weeks.
Period: Overall Study
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Started | 7443
Completed | 7443
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients enrolled, registered and received at least one dose were included in the treated set.
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7443
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated set (TS): All patients enrolled, registered and received at least one dose were included in the treated set.
  Years | 65.07 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated set (TS): All patients enrolled, registered and received at least one dose were included in the treated set.
  Participants
    Female | 2349
    Male | 5094
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success After Approximately 6 Weeks.
Description: The therapeutic success was defined as a minimum of 10- point increase in the Physical Functioning (PF-10) score between visit 1 (baseline visit at the start of the study) and visit 2 (final visit approximately 6 weeks after visit 1), having approximately time period of 6 weeks between the evaluated questionnaires. PF-10 score measures changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients.
Time Frame: Approximately 6 weeks
Population: Full analysis set (FAS): All patients who received treatment with Spiolto® Respimat® and had visits 1 and 2 documented as well as filled in all questionnaires were included in the full analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Percentage of participants (%) | 67.76 [66.67 to 68.84]

2. Secondary Outcome: Change in the Physical Functioning (PF-10) Score From Baseline (visit1) to Approximately 6 Weeks (visit2)
Description: Change in PF-10 score was determined by taking into account the individual change of each patient between visit 1 and visit 2. The PF-10 used for assessing the primary outcome is a sub-domain of the validated Short Form (SF)-36 quality of life questionnaire and consists of 10 questions evaluating the experienced restrictions while conducting usual activities. Each question of the PF-10 may be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3, respectively. The scores will be summed up between 10 and 30. The final sum of the individual scores was standardized to a range of 0 to 100 using the formula: 100*(sum-10)/20. The lower the score the more disability. The higher the score the less disability. If less than half of the scale items were missing, missing values were replaced with the mean of the other values. If half or more than half was missing, no score was calculated.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Score on scale | 16.62 (17.87)

3. Secondary Outcome: General Condition of the Patients Evaluated by the Physician, (Physician's Global Evaluation (PGE) Score) at Baseline (visit1) and Approximately 6 Weeks (visit2).
Description: This outcome measures general condition of the patient evaluated by the physician (PGE score) at visit 1 (baseline visit at the start of the study) and visit 2 (final visit approximately 6 weeks after visit 1) evaluated on an 8-point scale with the scores "Poor (1,2)", "Satisfactory (3, 4)", "Good (5, 6)" and "Excellent (7, 8)". More the score, the better is the general condition of patient.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Participants
  Score 1 at visit 1 | 96
  Score 2 at visit 1 | 754
  Score 3 at visit 1 | 1907
  Score 4 at visit 1 | 2159
  Score 5 at visit 1 | 1317
  Score 6 at visit 1 | 743
  Score 7 at visit 1 | 203
  Score 8 at visit 1 | 39
  Score 1 at visit 2 | 0
  Score 2 at visit 2 | 53
  Score 3 at visit 2 | 261
  Score 4 at visit 2 | 887
  Score 5 at visit 2 | 1772
  Score 6 at visit 2 | 2458
  Score 7 at visit 2 | 1451
  Score 8 at visit 2 | 335

4. Secondary Outcome: Patient's Overall Satisfaction With Treatment Spiolto® Respimat® at Visit 2 (Approximately 6 Weeks)
Description: At visit 2 patients were asked for their overall satisfaction with the Spiolto® Respimat® device. The patients were given range of responses from very satisfied to very dissatisfied and responses were recorded including unanswered cases.
Time Frame: Approximately 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Participants
  Very satisfied | 2847
  Satisfied | 2998
  Rather satisfied | 890
  Neither satisfied nor dissatisfied | 307
  Rather dissatisfied | 93
  Dissatisfied | 52
  Very dissatisfied | 26
  Not answered | 5

5. Secondary Outcome: Patient's Satisfaction With Inhaling From Device Spiolto® Respimat® at Visit 2 (Approximately 6 Weeks)
Description: At visit 2 patients were asked how satisfied they were with inhaling from the Spiolto® Respimat® device. The patients were given range of responses from very satisfied to very dissatisfied and responses were recorded including unanswered cases.
Time Frame: Approximately 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Participants
  Very satisfied | 3143
  Satisfied | 3021
  Rather satisfied | 716
  Neither satisfied nor dissatisfied | 228
  Rather dissatisfied | 48
  Dissatisfied | 34
  Very dissatisfied | 11
  Not answered | 17

6. Secondary Outcome: Patient's Satisfaction With Handling Inhalation Device Spiolto® Respimat® at Visit 2 (Approximately 6 Weeks)
Description: At visit 2 patients were asked how satisfied they were with handling the Spiolto® Respimat® device. The patients were given range of responses from very satisfied to very dissatisfied and responses were recorded including unanswered cases.
Time Frame: Approximately 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
Number analyzed (Participants) | 7218
Participants
  Very satisfied | 3086
  Satisfied | 2988
  Rather satisfied | 794
  Neither satisfied nor dissatisfied | 239
  Rather dissatisfied | 55
  Dissatisfied | 30
  Very dissatisfied | 9
  Not answered | 17

ADVERSE EVENTS:
Time Frame: From first dose adminstration until 21 days after permanently discontinuation of therapy or end of the study.
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Analysis of adverse events were done on Treated set, which includes all patients enrolled, registered and received at least one dose.
Arm/Group | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram
All-Cause Mortality (participants affected / at risk) | 4/7443
Serious Adverse Events (participants affected / at risk) | 5/7443
Other Adverse Events (participants affected / at risk) | 0/7443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® Respimat® 2.5 Microgram/ 2.5 Microgram (N=7443)
Atrial fibrillation (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
The impact and the interpretation of this data are limited due to the non-interventional study concept. No objective assessment was performed. It might be considered that patients may get used to limited activity and overrate their baseline activity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02719639/SAP_000.pdf
  • Study Protocol (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT02719639/Prot_001.pdf